CLINICAL TRIAL: NCT00908492
Title: Pilot Study of the Environmental Skill Building Program for Dementia Caregivers
Brief Title: Supporting Caregivers of Persons With Dementia: A Pilot Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Principal Investigator, Lori Letts, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC1050
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Randomized control trial; Dementia caregivers; Occupational Therapy; Caregivers
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Control (Active Comparator)
  Interventions: Behavioral: Education Control
- Environmental Skill Building (Experimental)
  Interventions: Behavioral: Environmental Skill Building

INTERVENTIONS:
Behavioral: Education Control — Caregiver participants are provided with information about caregiver stress and discuss it individually with an interventionist who visits the home. The control intervention involves 5 visits over 6 months.
  Arms: Education Control
Behavioral: Environmental Skill Building — The ESP intervention addresses home modifications and training in their use, instruction in strategies of problem-solving, energy conservation, safe task performance, fall recovery techniques, and balance and muscle strength training. Intervention is individualized for target areas identified in the initial client assessment and caregiver interview. The intervention involves using a problem solving approach and client-centred focus and the intervention assessment tools are individualized measures which determine the goals identified by the caregiver. It involves 5 visits over 6 months.
  Arms: Environmental Skill Building

SUMMARY:
The purpose of this study is to pilot the home Environmental Skill-Building Program (ESP) and an educational control intervention with persons with dementia and their caregivers (n=40) in preparation for a larger double-blind randomized controlled trial. Caregivers of persons with dementia often deal with difficult behaviors. The ESP is an occupational therapy intervention that helps caregivers adapt to their environment and build care-giving skills. The areas addressed include changes to the home set-up, adaptive equipment, instruction in strategies of problem-solving, energy conservation, safe task performance, and fall recovery techniques. A trial is needed with methodological rigor and to determine if the intervention is feasible in the Canadian health care system. Results will contribute to understanding how caregivers and people with dementia can be supported in their home environments.

ELIGIBILITY:
Inclusion Criteria:

* The caregiver must be the primary caregiver
* Caregiver reports that the care recipient has at least one limitation in basic activities of daily living (ADL) or two dependencies in instrumental activities of daily living (IADLs)
* The caregiver must:

  * provide at least 2 hours of care per day
  * be caregiving for at least 6 months and
  * be at least 21 years of age
* The care recipients need to have a diagnosis of dementia

Exclusion Criteria:

* Caregiver:

  * does not live with the care recipient
  * has poor health (undergoing treatments for cancer, hospitalized more than three times in past year)
  * planning to place care recipient in long term care within the next year
* Care recipients who are confined to bed most of the day or are minimally-responsive to touch or the environment are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Revised Memory and Behavior Problem Checklist | 0, 6, 9 months

SECONDARY OUTCOMES:
Disability Assessment for Dementia | 0, 6, 9 months
Number of caregiving assistance hours | 0, 6, 9 months
Short Zarit Burden Interview | 0, 6, 9 months
Task Management Strategy Index | 0, 6, 9 months
Perceived Change Scale | 0, 6, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Letts, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada